CLINICAL TRIAL: NCT01392443
Title: A Multi-national Open-label Phase II Study of the JAK Inhibitor INC424 in Patients With Primary Myelofibrosis, Post-polycythemia Vera Myelofibrosis or Post-essential Thrombocythemia Myelofibrosis
Brief Title: Asian Phase II Study of INC424 in Patients With Primary Myelofibrosis (MF), Post-PV MF or Post-ET MF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424A2202
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Results first posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Primary Myelofibrosis (MF); Post-Polycythemia Vera (PV) MF; Post-Essential Thrombocythemia (ET) MF
Keywords: Primary Myelofibrosis (MF); Post-Polycythemia Vera (PV) MF; Post-Essential Thrombocythemia (ET) MF; post-PV MF; post-ET MF; INC424; Ruxolitinib; Myelofibrosis; MF
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): Ruxolitinib was taken twice daily, unless instructed. Starting dose 15 mg BID for patients with baseline platelet count of 100,000/μL to 200,000/μL (inclusive) or 20 mg BID for those with baseline platelet count >200,000/μL (approximately 12 hours apart: morning and night), increased or decreased per standardized dosing paradigm.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — INC424 Tablet for oral use, provided in 5 mg bottles. The dosage strength was 5 mg/tablet INC424 phosphate (free base equivalent).
  Other Names: INC424

SUMMARY:
The objective of this study was to determine the efficacy of INC424 as assessed by reduction in spleen volume in patients with primary myelofibrosis (MF), post-polycythemia vera (PV) MF, or post-essential thrombocythemia (ET) MF. The safety and tolerability of INC424 and the effects of INC424 on patient reported outcomes and the duration of response as assessed by reduction in spleen volume was also assessed.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Diagnosis of primary myelofibrosis (MF), post-polycythemia vera (PV) MF, or post-essential thrombocythemia (ET) MF
3. Enlarged spleen, measuring 5 cm or greater from the costal margin
4. Must have two or more of the following risk factors:

   1. Over 65 years old
   2. Have the following symptoms often associated with MF: loss of weight, fever, night sweats
   3. Have a low red blood cell count (anemia - hemoglobin < 10 g/dL)
   4. Have a high white blood cell count (history of white blood cell count > 25,000/uL)
   5. Have high circulating blasts (> or = 1%) as measured by blood tests
5. Should have circulating blasts <10% (as measured by blood tests)
6. Should be capable of self-care
7. Should have adequate bone marrow reserve
8. Should not have the option of stem cell transplantation
9. Should discontinue any prior or ongoing treatment for myelofibrosis prior to entering the study
10. Had no prior treatment with another JAK inhibitor

Exclusion Criteria:

1. Does not have adequate liver or kidney function (as measured by blood tests)
2. Has an active infection (bacterial, viral, etc.)
3. Has active hepatitis A, B, or C or positive for HIV
4. Has another cancer that needs active intervention
5. Had a history of bleeding disorder
6. Had a history of very low platelet counts (as measured by blood tests) not related to treatment of MF
7. Had radiation of the spleen within 1 year of joining the study
8. Does not have adequate heart function
9. Sufficient time has elapsed between stopping previous treatment for MF and joining the study
10. Females who are pregnant or breast-feeding
11. Not able to sign informed consent
12. Has any other active medical conditions that the doctor deems may compromise your safety or ability to join in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-10-14 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- China (10):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Shanghai
- Japan (8):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- South Korea (3):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Seoul
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Jin J, Du X, Zhou DB, Li JM, Li JY, Hou M, Liu T, Wu DP, Hu Y, Xiao ZJ. [Efficacy and safety of JAK inhibitor ruxolitinib in Chinese patients with myelofibrosis: results of a 1-year follow-up of A2202]. Zhonghua Xue Ye Xue Za Zhi. 2016 Oct 14;37(10):858-863. doi: 10.3760/cma.j.issn.0253-2727.2016.10.007. Chinese. PMID 27801315

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 110 patients were planned, 120 patients were enrolled and analyzed.
Period: Overall Study
Arm/Group | Ruxolitinib
Started | 120
Completed (Completed = End of Treatment) | 52
Not Completed | 68
Not completed — Disease progression | 30
Not completed — Adverse Event | 24
Not completed — Death | 7
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): comprised of all patients who received at least one dose of ruxolitinib.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.0 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 58
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 30
  Korean | 17
  Chinese | 63
  Taiwanese | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 35% Reduction in Spleen Volume From Baseline at Week 24
Description: The primary measure of spleen size was by MRI. MRIs were performed with a body coil because the objective was to measure organ volume only, not to assess for lesions. MRIs were performed by local radiologists who were instructed not to provide a quantitative measure of spleen volume, but could provide a qualitative assessment such as enlarged, smaller, larger, etc. The scans from an individual patient were to be read by a central reader upon transfer from the site radiologist.
Time Frame: 24 weeks
Population: Full Analysis Set (FAS): comprised of all patients who received at least one dose of ruxolitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 120
Participants | 38
Statistical Analysis 1: Comparison: Ruxolitinib; Test type: Other; p = 0.0007, single-sample biniminal test

2. Secondary Outcome: Percentage of Participants With at Least 35% Reduction in Spleen Volume From Baseline at Each Scheduled Time Point - Best Response
Description: The best response rate was defined as the proportion of patients achieving a ≥ 35% reduction in spleen volume from baseline at any post-baseline assessment. The best response rate was estimated with an associated 95% confidence interval.
Time Frame: Weeks 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, at any time point
Population: Full Analysis Set (FAS): comprised of all patients who received at least one dose of ruxolitinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 120
Percentage of participants
  Week 24 | 35.8 [27.3 to 44.4]
  Week 36 | 40.0 [31.2 to 48.8]
  Week 48 | 44.2 [35.3 to 53.1]
  Week 72 | 44.2 [35.3 to 53.1]
  Week 96 | 45.8 [36.9 to 54.7]
  Week 120 | 45.8 [36.9 to 54.7]
  Week 144 | 46.7 [37.7 to 55.6]
  Week 168 | 47.5 [38.6 to 56.4]
  Week 192 | 47.5 [38.6 to 56.4]
  Week 216 | 47.5 [38.6 to 56.4]
  Week 240 | 47.5 [38.6 to 56.4]
  at any time point | 47.5 [38.6 to 56.4]

3. Secondary Outcome: Kaplan Meier Estimates of Duration of Response of at Least ≥ 35% Reduction From Baseline in Spleen Volume Per Kaplan Meier Estimates
Description: For patients who had at least one ≥ 35% reduction in spleen volume from baseline at postbaseline, the duration of response was calculated. The start date of the duration was defined as the first spleen volume measurement that was ≥ 35% reduction from baseline, and the end date of the response duration was defined as the earliest of the following: death, A ≥ 25% increase in spleen volume by MRI (or CT in applicable patients) compared to baseline, Splenic irradiation, Leukemic transformation as defined by a bone marrow or a peripheral blood blast count of ≥ 20%, Splenectomy. Duration of response is calculated only for participants who achieved at least one measured >= 35% reduction in spleen volume at any time.
Time Frame: Weeks 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240
Population: Full Analysis Set (FAS): comprised of all patients who received at least one dose of ruxolitinib.
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 120
weeks
  12 weeks | 1.00 [1.00 to 1.00]
  24 weeks | 0.96 [0.86 to 0.99]
  36 weeks | 0.96 [0.86 to 0.99]
  48 weeks | 0.93 [0.82 to 0.97]
  60 weeks | 0.93 [0.82 to 0.97]
  72 weeks | 0.91 [0.79 to 0.96]
  84 weeks | 0.89 [0.77 to 0.95]
  96 weeks | 0.89 [0.77 to 0.95]
  120 weeks | 0.89 [0.77 to 0.95]
  144 weeks | 0.85 [0.71 to 0.93]
  168 weeks | 0.79 [0.62 to 0.89]
  192 weeks | 0.75 [0.57 to 0.86]
  216 weeks | 0.75 [0.57 to 0.86]
  240 weeks | NA [NA to NA] — DOR calculated with 1 measured >= 35% reduction in spleen volume at any time - not reached for this time point.

4. Secondary Outcome: Change in EORTC QLQ-C30 Scores From Baseline in at Week 24
Description: Patient reported outcomes regarding the impact of MF on patients were assessed using the EORTC QLQ-C30. Data from the EORTC QLQ-C30 questionnaire was analyzed using the standardized scores. There were 2 categories to this scale: Functional/QOL scale and Symptom and Other items scale. For each sub-scale, the raw scores were standardized in order to obtain scores ranging from 0 to 100. For Functional/QOL subscales: a higher score represents a higher/better level of functioning. For Symptoms and Other items subscales: a higher score represents worse level of symptoms. The absolute change from baseline was calculated for each scale and summarized descriptively by scheduled visit.
Time Frame: Baseline, Week 24
Population: Full Analysis Set (FAS): comprised of all patients who received at least one dose of ruxolitinib.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 120
scores on a scale
  Func./QOL scales: Global Health Status/QOL: number analyzed (Participants) | 101
  Func./QOL scales: Global Health Status/QOL | 5.2 (22.04)
  Func./QOL scales: Physical Functioning: number analyzed (Participants) | 101
  Func./QOL scales: Physical Functioning | 0.6 (14.70)
  Func./QOL scales:Role Functioning: number analyzed (Participants) | 101
  Func./QOL scales:Role Functioning | -0.2 (21.54)
  Func./QOL scales: Emotional Functioning: number analyzed (Participants) | 101
  Func./QOL scales: Emotional Functioning | 1.9 (14.14)
  Func./QOL scales: Cognitive Functioning: number analyzed (Participants) | 101
  Func./QOL scales: Cognitive Functioning | -4.0 (18.43)
  Func./QOL scales: Social Functioning: number analyzed (Participants) | 101
  Func./QOL scales: Social Functioning | 0.2 (21.41)
  Symptom and Other items: Fatigue: number analyzed (Participants) | 101
  Symptom and Other items: Fatigue | -1.3 (20.32)
  Symptom & Other items: Nausea and Vomiting: number analyzed (Participants) | 101
  Symptom & Other items: Nausea and Vomiting | 0.0 (9.43)
  Symptom and Other items: Pain: number analyzed (Participants) | 101
  Symptom and Other items: Pain | -1.8 (18.99)
  Symptom and Other items: Dyspnea: number analyzed (Participants) | 101
  Symptom and Other items: Dyspnea | 2.3 (25.93)
  Symptom and Other items: Insomnia: number analyzed (Participants) | 101
  Symptom and Other items: Insomnia | -2.0 (30.12)
  Symptom and Other items: Appetite Loss: number analyzed (Participants) | 101
  Symptom and Other items: Appetite Loss | -6.3 (25.26)
  Symptom and Other items: Constipation: number analyzed (Participants) | 101
  Symptom and Other items: Constipation | 4.6 (20.02)
  Symptom and Other items: Diarrhea: number analyzed (Participants) | 101
  Symptom and Other items: Diarrhea | 1.7 (23.75)
  Symptom & Other items: Fin. difficulties: number analyzed (Participants) | 101
  Symptom & Other items: Fin. difficulties | -2.0 (23.49)

5. Secondary Outcome: Change in Total Symptom Score From Baseline at Week 24 as Measured by Seven-day Modified MFSAF v2.0
Description: The Seven-day modified MFSAF v2.0 is a 7-item PRO instrument based on the modified MFSAF v2.0 diary administered at specified visits. Symptoms of myelofibrosis (MF) were assessed using this instrument & included filling up quickly/early satiety, abdominal discomfort, pain under the ribs, night sweats, itching, bone/muscle pain & inactivity. The first 6 items assessed MF symptom severity at its worst as recalled & the seventh captured MF-related inactivity in the 7 days prior to the clinic visit assessment. All 7 items asked subjects to record their answers on an 11-point numeric rating scale (NRS) (0=Absent, 10=Worst Imaginable). The first 6 items of the instrument focus on MF symptoms & are summed to create a Total Symptom score, defined as the sum of the 6 individual symptom scores other than the inactivity score (each with 0-10 point scale) collected on the same week. The total symptom scale ranges from 0 -60 where higher score indicates a worse level of the condition.
Time Frame: Baseline, Week 24
Population: Full Analysis Set (FAS): comprised of all patients who received at least one dose of ruxolitinib.
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 120
scores on a scale | -5.0 [-27 to 21]

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse Events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to 240 weeks.
Arm/Group | Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 13/120
Serious Adverse Events (participants affected / at risk) | 60/120
Other Adverse Events (participants affected / at risk) | 117/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=120)
Anaemia (Blood and lymphatic system disorders) | 5
Coagulopathy (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 3
Cardiac failure acute (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Disuse syndrome (General disorders) | 1
Pyrexia (General disorders) | 8
Sudden death (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Abdominal infection (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Enteritis infectious (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 6
Infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 9
Pneumonia bacterial (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Soft tissue infection (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Bone contusion (Injury, poisoning and procedural complications) | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Bilirubin conjugated increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Langerhans' cell histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Calculus bladder (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1
Aortic dissection (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Peripheral embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=120)
Anaemia (Blood and lymphatic system disorders) | 87
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 34
Abdominal distension (Gastrointestinal disorders) | 25
Abdominal pain (Gastrointestinal disorders) | 14
Abdominal pain upper (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 21
Diarrhoea (Gastrointestinal disorders) | 42
Dyspepsia (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 9
Stomatitis (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 9
Asthenia (General disorders) | 19
Fatigue (General disorders) | 12
Malaise (General disorders) | 8
Oedema peripheral (General disorders) | 20
Pain (General disorders) | 11
Pyrexia (General disorders) | 26
Herpes zoster (Infections and infestations) | 18
Nasopharyngitis (Infections and infestations) | 24
Upper respiratory tract infection (Infections and infestations) | 38
Alanine aminotransferase increased (Investigations) | 26
Aspartate aminotransferase increased (Investigations) | 23
Blood bilirubin increased (Investigations) | 9
Blood creatinine increased (Investigations) | 10
Blood iron increased (Investigations) | 7
Blood urea increased (Investigations) | 8
C-reactive protein increased (Investigations) | 11
Gamma-glutamyltransferase increased (Investigations) | 19
Lymphocyte count decreased (Investigations) | 11
Neutrophil count decreased (Investigations) | 11
Platelet count decreased (Investigations) | 44
Weight increased (Investigations) | 15
White blood cell count decreased (Investigations) | 8
Decreased appetite (Metabolism and nutrition disorders) | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 17
Hypocalcaemia (Metabolism and nutrition disorders) | 9
Iron overload (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 10
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 16
Insomnia (Psychiatric disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 31
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9
Night sweats (Skin and subcutaneous tissue disorders) | 13
Pruritus (Skin and subcutaneous tissue disorders) | 15
Hypertension (Vascular disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2011-04-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT01392443/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT01392443/SAP_001.pdf